CLINICAL TRIAL: NCT00188318
Title: A Phase II Study of Hyperfractionated Accelerated Radiotherapy Delivered With Integrated Neck Surgery for Node-positive Cases in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Hardwins - Squamous Cell Carcinoma Head & Neck (Surgery/RT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0557-C
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell

ARMS (1):
- Hyperfractionated Accelerated Radiotherapy (Experimental): Hypofractionated Accelerated Radiotherapy with integrated neck surgery
  Interventions: Procedure: hyperfractionated accelerated radiotherapy

INTERVENTIONS:
Procedure: hyperfractionated accelerated radiotherapy

SUMMARY:
This study is examining the effects of increasing the dose of radiation given to treat head and neck cancer. Radiation doses to the primary cancer are higher than usually given; lymph glands of the neck will also be treated at a lower dose. Surgery on the lymph glands my be necessary in the future. Radiation treatments given in small fractions twice a day allows a higher dose to be delivered than if the treatment was given once a day. This study will enroll patients at three sequential increasing dose levels. Approximately 40 patients will be enrolled at each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma
* Larynx & pharynx (except Nasopharyngeal carcinoma)
* Stage III & IV, but any stage hypopharynx
* Informed Consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 1998-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Toxicities as per CTCAE | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: John Waldron, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada